CLINICAL TRIAL: NCT06796829
Title: Nutritional Status of Pregnant Women Following Bariatric Surgery
Acronym: NEWBIE
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Maxima Medical Center (Other); Gelderse Vallei Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1267
Record Dates: First submitted 2025-01-02; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions; Pregnancy; Metabolic Surgery
Keywords: Nutrient status; Nutritional supplementation; Metabolic bariatric surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to learn more about nutrient status during pregnancy after bariatric surgery. All pregnant women older than 18 years who underwent bariatric surgery and sought obstetric care within one of the participating hospitals were included and followed up until 2 months post-partum.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Medical history of metabolic bariatric surgery (Roux-en-Y gastric bypass or sleeve gastrectomy)

Exclusion Criteria:

* Elective termination of pregnancy
* Multiple pregnancy
* Metabolic bariatric procedures other than Roux-en-Y gastric bypass or sleeve gastrectomy
* Reversal of the bariatric procedure
* Malnutrition due to other causes (e.g., malignancy, alcoholism)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study on pregnancy. Therefore limited to female sex at birth.
Study Population: All pregnant women older than 18 years with a medical history of metabolic bariatric surgery presenting at the obesity or antenatal clinic at one of the participating centers were eligible for recruitment. Participants were preferably included before 12 weeks of pregnancy and followed up until 2 months post-partum.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Nutrient status during pregnancy | Nutrient status was preferably assessed at 4 occasions: During trimester 1 (week 1-12), trimester 2 (week 13-26), trimester 3 (week 27-42) and at 2 months post-partum.
  Nutrient deficiencies during each trimester of pregnancy. Nutrients of primary interest include ferritin, folic acid, vitamin A-D-B12 and albumin.

SECONDARY OUTCOMES:
Neonatal birth weight | Directly after delivery/birth
  Neonatal birth weight, weight-for-age percentile and classification of small-for-gestational age.
Gestational weight gain | From the beginning of pregnancy (max 3 months before conception until 1 month after conception) until date of delivery (max 2 weeks before event)
  Gestational weight gain in kg and classification of weight gain according to IOM recommendations.

OTHER OUTCOMES:
Use of supplementation | At trimester 1 (week 1-12), trimester 2 (week 13-26), trimester 3 (week 27-42) and at 2 months post-partum.
  Self-reported use of (multivitamin) supplementation
Surgery characteristics | At estimated date of conception (first day of last menstrual period + 14 days)
  Type of bariatric procedure and time from surgery to conception
Pregnancy outcomes | From the estimated date of conception (first day of last menstrual period + 14 days) until date of delivery
  Incidence of pregnancy complications including spontaneous abortion, preterm birth, gestational diabetes mellitus, hypertensive disorders, hyperemesis gravidarum, internal herniation, birth defects, NICU admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate/Vitalys, Elst, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heusschen L, Berendsen AAM, van Bon AC, van Laar JOEH, Krabbendam I, Hazebroek EJ. Nutrient Status and Supplement Use During Pregnancy Following Metabolic Bariatric Surgery: A Multicenter Observational Cohort Study. Obes Surg. 2024 Oct;34(10):3608-3618. doi: 10.1007/s11695-024-07446-4. Epub 2024 Aug 14. PMID 39141187